CLINICAL TRIAL: NCT02772731
Title: A Multicenter Randomized Controlled Trial of Routine Shave Margins vs. Standard Partial Mastectomy in Breast Cancer Patients
Brief Title: Shave Margins vs. Standard Partial Mastectomy in Breast Cancer Patients
Acronym: SHAVE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1602017205
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shave Margin (Experimental): After partial mastectomy, patients will be subject to intraoperative randomization to the shave margin group where additional tissue will be resected.
  Interventions: Procedure: Partial mastectomy plus additional Shave Margin
- No Shave Margin (Active Comparator): After partial mastectomy, patients will be subject to intraoperative randomization to the no shave margin group, where after initial surgery, no further tissue will be removed.
  Interventions: Procedure: Partial mastectomy

INTERVENTIONS:
Procedure: Partial mastectomy plus additional Shave Margin — For the shave group, additional superior, inferior, medial and lateral margins will be removed, oriented, and sent for pathologic evaluation at the local site. Resection of additional anterior and posterior margins will be left to surgeon discretion, as this will depend on if skin or fascia was taken. All surgeons participating in the study will be educated on the expectation of what is considered a "shave margin". A shave margin is defined as an additional segment of breast tissue taken from each of the superior, inferior, medial, and lateral aspects of the cavity, such that the entire circumference of the cavity is re-excised following this procedure. Orientation of each shaved margin will be done to mark the true margin.
  Arms: Shave Margin
Procedure: Partial mastectomy — Surgeons will be instructed to close after partial mastectomy with no further excision.
  Arms: No Shave Margin

SUMMARY:
Breast cancer is the most common malignancy affecting women in the US. Surgical management is the mainstay of therapy, and in general consists of resection of the primary tumor with either a partial mastectomy (aka "lumpectomy") or a total mastectomy.

The investigators hypothesize that routine shave margins during partial mastectomy will significantly reduce positive margin rate. A positive margin means that cancerous cells were detected at the edge of the excised area. This generally mandates a return to the operating room for re-excision.

DETAILED DESCRIPTION:
Some authors have investigated, in a retrospective fashion, the use of routine shave margins, where surgeons routinely take additional margins at the time of the initial partial mastectomy as a means of obtaining negative margins. While these retrospective studies have found that positive margin rates declined using this technique, opponents to this technique wonder if this truly results in a higher negative margin rate without compromising cosmesis or increasing tissue volume removed. As these studies were retrospective, it was possible that the initial resection was smaller than what those who do not routinely take shave margins would resect. No one had evaluated the impact of further resection on operative time, nor in a blinded fashion, evaluated cosmesis. Further, there had yet to be a prospective study to evaluate the impact of this on local recurrence rates. Hence, the investigators performed a prospective randomized controlled trial of this technique at Yale. The data from this study, published in the New England Journal of Medicine, found that the technique cut positive margin and re-excision rates in half. Some wondered, however, about the external generalizability of these findings, particularly in non-academic settings. Hence, a multicenter trial to validate these findings is warranted.

ELIGIBILITY:
Inclusion Criteria

1. Breast cancer, stage 0-3, deemed a surgically appropriate candidate for partial mastectomy with planned procedure for the same
2. Women ≥ 18 years of age
3. Ability to understand and the willingness to sign a written informed consent document.

Exlusion Criteria

1. Total mastectomy
2. Known metastatic disease
3. Bilateral synchronous breast cancer
4. Multicentric cancers requiring double lumpectomy
5. Previous history of breast cancer (even in the other breast)
6. Patients receiving Intraoperative radiation therapy (IORT)
7. Patients who had excisional biopsy for diagnosis of their cancer (I.e., instead of a core biopsy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06 (Actual); Study Completion 2024-11 (Actual)

PRIMARY OUTCOMES:
Positive margin rate | immediately after surgery
  The effect is positive margin rate post-surgery as measured by local pathological reports. Positive margins were defined as tumor touching the edge of the specimen that was removed in patients with invasive cancer and tumor that was within 2 mm of the edge of the specimen removed in those with ductal carcinoma in situ.

SECONDARY OUTCOMES:
local recurrence rates | up to 5 years
  Patients will be assessed for local recurrence based on physical examination, mammography, and follow up phone calls. This is a composite score with only one outcome and only one unit (respondents). A positive results from any of these methods indicates recurrence.
patient perceived cosmesis | 1 year post-op
  Subjects will be asked their perception of physical appearance: poor, fair, good, or excellent.
patient perceived cosmesis | 5 years post-op
  Subjects will be asked their perception of physical appearance: poor, fair, good, or excellent.
volume of tissue resected | immediately after tissue resection
  based on the sum of the volumes of tissue excised as found in the gross description of the specimens on the pathology report.
Quality of Life assessment | 1 year post-op about the last seven days
  Quality of Life Questionnaire measures quality of life over the past 7 days and includes 75 questions that are answered on a Likert scale. Questions assess physical, social, emotional and functional well-being in addition to cosmetic and physical appearance and questions regarding the surgery. Higher scores indicate a higher quality of life.
Quality of Life assessment | 5 years post-op about the last seven days
  Quality of Life Questionnaire measures quality of life over the past 7 days and includes 75 questions that are answered on a Likert scale. Questions assess physical, social, emotional and functional well-being in addition to cosmetic and physical appearance and questions regarding the surgery. Higher scores indicate a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Anees Chagpar, MD, Principal Investigator — Yale University
Locations (9):
- United States (9):
  - Loma Linda University Cancer Center, Loma Linda, California
  - Watson Clinic Cancer and Research Center, Lakeland, Florida
  - William Beaumont Hospital, Troy, Michigan
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Doctors Hospital at Renaissance, Edinburg, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chagpar AB, Killelea BK, Tsangaris TN, Butler M, Stavris K, Li F, Yao X, Bossuyt V, Harigopal M, Lannin DR, Pusztai L, Horowitz NR. A Randomized, Controlled Trial of Cavity Shave Margins in Breast Cancer. N Engl J Med. 2015 Aug 6;373(6):503-10. doi: 10.1056/NEJMoa1504473. Epub 2015 May 30. PMID 26028131